CLINICAL TRIAL: NCT04475445
Title: Fluoroscopic Guided Interlaminar Epidural Versus Ultrasound Guided Transforaminal Epidural in the Treatment of Unilateral Cervicobrachialgia : a Randomized Controlled Trial
Brief Title: Fluoroscopic Guided Interlaminar Epidural Versus Ultrasound Guided Transforaminal Epidural in the Treatment of Unilateral Cervicobrachialgia.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE/20-04-08
Record Dates: First submitted 2020-07-02; First posted 2020-07-17 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Cervicobrachial Neuralgia
Keywords: Neuropathic Cervicobrachial; Ultrasound-guided transforaminal infiltration; Cervical Interlaminar epidural infiltration; Cervical Chronic Pain
MeSH Terms: conditions — Brachial Plexus Neuritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound guided transforaminal epidural steroid injection (Experimental)
  Interventions: Other: Ultrasound-guided transforaminal epidural steroid injection
- Interlaminar epidural steroid injection (Experimental)
  Interventions: Other: Interlaminar epidural steroid injection

INTERVENTIONS:
Other: Ultrasound-guided transforaminal epidural steroid injection — Ultrasound identification of the nerve root, fluoroscopic control of the position and injection of a mixture of 10 mg of dexamethasone and 20 mg of lidocaine.
  Arms: Ultrasound guided transforaminal epidural steroid injection
Other: Interlaminar epidural steroid injection — Fluoroscopic location of the epidural space C5C6 or C6C7, injection of a mixture of 10 mg of dexamethasone and 20 mg of lidocaine.
  Arms: Interlaminar epidural steroid injection

SUMMARY:
Chronic cervicobrachialgia is a public health problem. Epidural injections of corticosteroids and local anesthesics via transforaminal and interlaminar routes both have shown their potential in its treatment. The interlaminar approach offers the advantage of an epidural injection (i.e., direct contact with the nerve root in the epidural space). However, it requires fluoroscopy and can lead to potentially serious complications (compression of the nerve root, spinal cord injury...). The ultrasound-guided injection of corticosteroids via the transforaminal route, which offers the advantage of selectively targeting the symptomatic nerve root, may have the same therapeutic advantages as the interlaminar approach in decreasing unilateral cervicobrachial pain (i.e. a decrease in pain after infiltration) and reduce its risks.The aim of this study is to compare the efficacy of transforaminal vs interlaminar cervical corticosteroid injection.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status (ASA) I-III
* Chronic unilateral cervicobrachial pain
* Allowed Steroid infiltration

Exclusion Criteria:

* Pregnancy
* Lactation
* Allergy or intolerance to any of the drugs/materials used in this study,
* Participation in another interventional study
* Systemic anticoagulation,
* Infection at the puncture site
* Patient refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-07-30 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Score change at 30 minutes post infiltration when compared to baseline | up to 30 minutes
  Pain will be evaluated by Visual Analog Scale (VAS) before and 30 minutes after corticosteroid infiltration.
  Visual Analog pain score (scale = 0 no pain; 10= worst pain imaginable)

SECONDARY OUTCOMES:
Visual Analogue Score change at 1 month post infiltration when compared to baseline | up to 1 month
  Pain will be evaluated by Visual Analog Scale (VAS) before and 1 month after corticosteroid infiltration.
  Visual Analog pain score (scale = 0 no pain; 10= worst pain imaginable)
Patient satisfaction during procedure | at the end of infiltration
  Pain will be evaluated by Satisfaction scale after procedure (0= unsatisfied, 5= very satisfied)
Neck disability index (NDI) score (questionnaire) | up to 1 month
  Neck disability index (NDI) score will be calculated before, 30 minutes and 1 month after corticosteroid infiltration
  The NDI is a standard instrument for measuring self-rated disability due to neck pain.
  Each of the 10 items is scored from 0 - 5. The maximum score is therefore 50. Points summed to a total score. The test can be interpreted as a raw score, with a maximum score of 50, Interpretation for scoring intervals : 0 - 4 = no disability; 5 - 14 = mild disability; 15 - 24 = moderate disability; 25 - 34 = severe disability, above 34 = complete disability.
Rate of Procedure failure | up to 30 minutes
  The procedure will be considered as a failure if the infiltration is not performed.
Incidence of Adverse effects (lipothymia, nausea, vomiting) | up to 1 month
Incidence of complications (stroke, hematoma, paralysis) | up to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Panayota Kapessidou, MD,PhD, Study Director — University Hospital Saint-Pierre (CHU Saint-Pierre), Université Libre de Bruxelles (ULB); Mohamed Ali Bali, MD, Principal Investigator — mohamed_bali@stpierre-bru.be
Locations (1):
- CHU Saint-Pierre, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaye AD, Manchikanti L, Abdi S, Atluri S, Bakshi S, Benyamin R, Boswell MV, Buenaventura R, Candido KD, Cordner HJ, Datta S, Doulatram G, Gharibo CG, Grami V, Gupta S, Jha S, Kaplan ED, Malla Y, Mann DP, Nampiaparampil DE, Racz G, Raj P, Rana MV, Sharma ML, Singh V, Soin A, Staats PS, Vallejo R, Wargo BW, Hirsch JA. Efficacy of Epidural Injections in Managing Chronic Spinal Pain: A Best Evidence Synthesis. Pain Physician. 2015 Nov;18(6):E939-1004. PMID 26606031
- [Background] Banik RK, Chen Chen CC. Spinal Epidural Hematoma after Interlaminar Cervical Epidural Steroid Injection. Anesthesiology. 2019 Dec;131(6):1342-1343. doi: 10.1097/ALN.0000000000002896. No abstract available. PMID 31365368
- [Background] Bush K, Mandegaran R, Robinson E, Zavareh A. The safety and efficiency of performing cervical transforaminal epidural steroid injections under fluoroscopic control on an ambulatory/outpatient basis. Eur Spine J. 2020 May;29(5):994-1000. doi: 10.1007/s00586-019-06147-2. Epub 2019 Sep 18. PMID 31535205
- [Background] Narouze SN, Vydyanathan A, Kapural L, Sessler DI, Mekhail N. Ultrasound-guided cervical selective nerve root block: a fluoroscopy-controlled feasibility study. Reg Anesth Pain Med. 2009 Jul-Aug;34(4):343-8. doi: 10.1097/AAP.0b013e3181ac7e5c. PMID 19574867